CLINICAL TRIAL: NCT00108563
Title: VISN 20 Prophylactic Treatment of IFN-Induced Depression in Hepatitis C
Brief Title: VISN 20: Prophylactic Treatment of Interferon-Induced Depression in Hepatitis C Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CLIN-012-02S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Hepatitis C; Depression
Keywords: Hepatitis C; Depression; Interferon-alpha; Citalopram; ribavirin; antidepressive agents
MeSH Terms: conditions — Hepatitis C; Depression | interventions — Citalopram

INTERVENTIONS:
Drug: Citalopram or Placebo

SUMMARY:
The purpose of this study is to learn more about the effects of interferon and ribavirin combination therapy in people with Hepatitis C. The specific aims are:

* To assess how often depressive symptoms occur in patients taking combination alpha interferon plus ribavirin or pegylated interferon plus ribavirin therapy for Hepatitis C, when depressive symptoms occur, and how severe the depressive symptoms are when they do occur;
* To identify potential predictors for the development of depressive symptoms;
* To identify if citalopram, an antidepressant medication, can prevent or lessen the severity of depressive symptoms brought about by interferon therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, age 18 or older
* Planning to receive any brand of pegylated interferon/ribavirin combination therapy for chronic HCV (hepatitis C virus)

Exclusion Criteria:

* Chronic liver disease other than chronic HCV
* Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy
* A history of organ transplantation
* Any known preexisting medical condition that could interfere with the patient's participation in the protocol, including: *active seizure disorders requiring medication; *history of major CNS (central nervous system) trauma (as suggested by accident or other event leading to loss of consciousness, personality changes, etc)
* Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids (e.g. oral or injection).
* Inability to read and write at a level sufficient to complete self-report forms
* History of significant non-compliance with medical treatments and appointments
* Patients currently, or within the last three months, on a full therapeutic dose of antidepressant medication, or a dose of other medication such that it may significantly affect depressive symptomatology
* Patients with active depression in the previous 3 months and/or those with BDI (Beck Depression Inventory)-II greater than or equal to 15 at the time of study entry.
* Patients with bipolar disorder or history of bipolar disorder
* Patients with active psychotic symptoms or diagnosis of schizophrenia in the previous 3 months
* Active substance abuse, such as alcohol (greater than 80 gm/day), IV (intravenous) drugs, and inhaled drugs. If the patient has a history of substance abuse, in order to be considered for inclusion into the protocol, the patient must have been in a sustained remission for at least 6 months
* Patients receiving opiate agonist therapy (e.g., methadone maintenance therapy) within the past year, unless a program of testing for continued substance abuse is initiated (testing at entry and then randomly at least every 2-3 months) and the patient is withdrawn from study for any violation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Portland, Oregon, United States